CLINICAL TRIAL: NCT03331185
Title: Dimensional Changes of Soft and Hard Tissues Following Alveolar Ridge Preservation: Freeze-dried Bone Allograft vs. L-PRF Clot Covered With d-PTFE Membrane: A Randomized Clinical Trial
Brief Title: Changes of Soft and Hard Tissues After Alveolar Ridge Preservation: Freeze-dried Bone Allograft vs. L-PRF Clot
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Jonathan Bouwer, Periodontal Resident, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017:125
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Alveolar Bone Loss; Tooth Loss
Keywords: Extraction; Alveolar Ridge Augmentation; Freeze Dried Bone Allograft; Leukocytic Platelet Rich Fibrin; Volumetric Changes; Dense Polytetrafluoroethylene Membrane
MeSH Terms: conditions — Alveolar Bone Loss; Tooth Loss

STUDY DESIGN:
Intervention Model Description: A prospective,randomized clinical trial will be conducted. The trial aims at obtaining information to determine which material would provide a superior clinical result, as well as reporting on patient related outcomes. 42 participants will be randomly assigned to two groups and a direct comparison will be made between the results obtained from the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Freeze Dried Bone Allograft (Active Comparator): Socket filled with Mineralized Cortical Freeze Dried Bone Allograft
  Interventions: Biological: Freeze Dried Bone Allograft
- L-PRF Clot (Experimental): Socket filled with L-PRF Clot
  Interventions: Biological: L-PRF clot

INTERVENTIONS:
Biological: Freeze Dried Bone Allograft — Human derived bone particles used in oral and periodontal grafting procedures
  Other Names: FDBA
  Arms: Freeze Dried Bone Allograft
Biological: L-PRF clot — L-PRF is a second-generation platelet rich plasma obtained from autologous blood and contains several different growth factors, platelets and leucocytes in a complex fibrin matrix to accelerate the healing of soft and hard tissues.
  Other Names: Leukocytic Platelet Rich Fibrin Clot
  Arms: L-PRF Clot

SUMMARY:
A Clinical Trial to study the effectiveness between two, tooth socket grafting materials namely, Freeze Dried Bone Allograft (human derived bone particles) and Leukocytic-Platelet Rich Fibrin (the patient's own centrifuged blood).

The purpose of this study is to compare the effects (good and bad) of Bone Allograft to Platelet Rich Fibrin to see which material would be the most effective in maintaining the volume of the gum and bone of the jaw during the healing phase as well as minimizing the amount of pain and/or swelling following tooth extraction.

DETAILED DESCRIPTION:
A prospective,randomized clinical trial will be conducted to determine whether L-PRF, compared to freeze dried bone allograft, will result in comparable volumetric shrinkage of the alveolar ridge and overlying keratinized tissue, following extraction of teeth and socket grafting.

This trial aims at obtaining information to determine which material would provide a superior clinical result, as well as reporting on patient related outcomes. The participants will be randomly assigned to two groups. The surgical procedure will be performed by one of five calibrated periodontal residents.

Patients will be followed for 2 weeks post-operatively by the same resident, to monitor the healing process and to assess for any complications.

Randomization will be achieved using a computerized randomization scheme and will be assigned to one of two groups and allocated by means of a sealed envelope opened on the day of surgery communicated to the surgeon during the surgery by a supervising faculty member. Participants will be block-randomized for each of the 5 operators for balance.

Anesthesia will be achieved and soft tissue measurements will be obtained using a periodontal probe. An atraumatic extraction technique will be performed to allow for minimal disturbance of the soft and hard tissue architecture.

The extraction socket walls are then assessed and any defects in socket measured with a periodontal probe. Group A: Full thickness mucoperiosteal pouch is created up to ~3mm apical of the bony crest of the socket with a periosteal elevator. The socket is incrementally filled with mineralized cortical freeze-dried bone allograft and condensed. Group B: Socket is pouched as in group A followed by venipuncture of the antecubital vein with 21G needle and collection of 4-6 vials (10ml each) of venous blood without any additive or anticoagulant. The vials are centrifuged for 12 minutes at 2700 rpm to form L-PRF clots. The socket is incrementally filled with the clots and condensed.

Following socket fill, both groups will have the grafts covered by dense polytetrafluoroethylene membrane. The membrane is trimmed and adapted with the borders tucked 2-3mm underneath the gingival tissues. Tissues, graft and membrane are stabilized with 5/0 PTFE sutures.

The patients will also receive a pain VAS questionnaire evaluating the post-operative pain 1 and 7 days following surgery. A CBCT with the radiographic stent will be taken within 72 hours of the surgery.

7 days post-op: Sutures will be removed if deemed suitable. The VAS questionnaire will be collected.

6 weeks post op: d-PTFE membrane will be retrieved and discarded using tissue forceps. Alginate impressions will be taken for a surgical guide.

11 weeks post op: Second CBCT will be taken with radiographic surgical stent. Images obtained will be used to analyze and compare the ridge dimensions to those obtained at baseline as well as for surgical implant planning.

12 weeks post op: Soft tissue measurement with periodontal probe and floss spanned over edentulous site from buccal to lingual mucogingival junction. Implant placement will be done per standard procedure. A 2.5mm diameter trephine drill will be used to harvest a bone core for histologic analysis. The bone core will be immediately submerged in a solution of 10% neutral buffered formalin. Osteotomies and implant placement will be done following the manufacturer's protocol. Depending on the buccal bone and soft tissue thickness, ancillary soft tissue augmentation, bone augmentation or combination of these procedures may be indicated. The patient will be followed up and referred to the restorative dentist as per standard procedure. Photographs will be taken at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with molars or premolars indicated for extraction.
* Patients that present with a post extraction class I and II socket (<30% bone loss on the buccal or lingual plate, measured from the most coronal aspect of intact bone to the most apical aspect of the defect divided by the measurement from the most apical aspect of the defect to the apex of the socket x 100).
* Patients presenting with the need for single extractions.
* Patients with general good health that does not have a condition contra-indicating routine dental treatment, extraction and implant placement.
* Patients that are compliant with the research protocol and methods.
* Patients that have read, understood and signed an informed consent form.

Exclusion Criteria:

* Extraction and ridge preservation indicated for teeth other than premolars and molars.
* Patients that present with a post extraction class III socket (>30% bone loss on the buccal or lingual plate, measured from the most coronal aspect of intact bone to the most apical aspect of the defect divided by the measurement from the most apical aspect of the defect to the apex of the socket x 100)
* Patients deemed eligible for immediate implant placement following extraction and intra-operative assessment by the attending supervisor.
* Patients that present with an oral-antral communication, post extraction.
* Patients that presents with the need for multiple, side by side extractions.
* Patients with coagulation disorders, on corticosteroids, uncontrolled diabetes mellitus, or any systemic disease where periodontal surgery is contraindicated and healing may be compromised.
* Pregnant and nursing women.
* Patients with any contact hypersensitivity to the related materials used in the study.
* Heavy tobacco users, >10 cigarettes per day.
* Patients unwilling to sign consent or follow the protocol of the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Cholakis, DDS, Study Director — University of Manitoba, Faculty of Graduate Studies, Periodontics
Locations (1):
- Graduate Periodontic Clinic - University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temmerman A, Vandessel J, Castro A, Jacobs R, Teughels W, Pinto N, Quirynen M. The use of leucocyte and platelet-rich fibrin in socket management and ridge preservation: a split-mouth, randomized, controlled clinical trial. J Clin Periodontol. 2016 Nov;43(11):990-999. doi: 10.1111/jcpe.12612. Epub 2016 Sep 21. PMID 27509214
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Walker CJ, Prihoda TJ, Mealey BL, Lasho DJ, Noujeim M, Huynh-Ba G. Evaluation of Healing at Molar Extraction Sites With and Without Ridge Preservation: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):241-249. doi: 10.1902/jop.2016.160445. Epub 2016 Oct 27. PMID 27788625
- [Background] Fernandez RF, Bucchi C, Navarro P, Beltran V, Borie E. Bone grafts utilized in dentistry: an analysis of patients' preferences. BMC Med Ethics. 2015 Oct 20;16(1):71. doi: 10.1186/s12910-015-0044-6. PMID 26486125
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Hauser F, Gaydarov N, Badoud I, Vazquez L, Bernard JP, Ammann P. Clinical and histological evaluation of postextraction platelet-rich fibrin socket filling: a prospective randomized controlled study. Implant Dent. 2013 Jun;22(3):295-303. doi: 10.1097/ID.0b013e3182906eb3. PMID 23644909
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part B: sinus floor elevation, alveolar ridge preservation and implant therapy. A systematic review. J Clin Periodontol. 2017 Feb;44(2):225-234. doi: 10.1111/jcpe.12658. Epub 2017 Jan 10. PMID 27891638
- [Background] MacBeth N, Trullenque-Eriksson A, Donos N, Mardas N. Hard and soft tissue changes following alveolar ridge preservation: a systematic review. Clin Oral Implants Res. 2017 Aug;28(8):982-1004. doi: 10.1111/clr.12911. Epub 2016 Jul 26. PMID 27458031
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.43 (12.92) | 63.33 (14.66) | 62.31 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 12 | 26
Buccolingual Ridge Width measured 1mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage that occurred during the healing phase
  Millimeters | 11.38 (2.4) | 11.28 (1.41) | 11.3 (1.8)
Buccolingual Ridge Width measured 3mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage that occurred during the healing phase
  Millimeters | 11.82 (2.37) | 12.20 (1.53) | 12 (1.9)
Buccolingual Ridge Width measured 5mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage that occurred during the healing phase
  Millimeters | 12.17 (2.49) | 12.47 (1.94) | 12.3 (2.2)
Thickness of buccal plate measured at 1mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage, of the buccal plate, that occurred during the healing phase
  Millimeters | 0.98 (0.5) | 0.89 (0.3) | 0.93 (0.4)
Thickness of buccal plate measured at 3mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage, of the buccal plate, that occurred during the healing phase
  Millimeters | 1.08 (0.8) | 1.31 (0.58) | 1.19 (0.69)
Thickness of buccal plate measured at 5mm from crest [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained will be compared to measurements taken at 11weeks to calculate the amount of horizontal shrinkage, of the buccal plate, that occurred during the healing phase
  Millimeters | 1.26 (0.98) | 1.50 (0.64) | 1.38 (0.8)
Buccolingual Keratinised Tissue Width [Mean (Standard Deviation); unit: Millimeters] — Baseline measurements obtained by measuring form the buccal to lingual mucogingival junction and compared to measurements taken at 12weeks to calculate loss/growth of keratinized tissue after healing.
  Millimeters | 15.25 (5.32) | 16.4 (4.39) | 15.8 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Overall Horizontal Change in Alveolar Ridge Width
Description: Calculated mean of post operative CBCT measurements of horizontal alveolar bone width changes following extraction and alveolar ridge preservation.
Time Frame: Difference reported on horizontal changes comparing CBCT analysis 11weeks after extraction and grafting compared to CBCT following extraction and grafting
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot
Number analyzed (Participants) | 14 | 12
Millimeters | -1.34 (0.38) | -2.21 (0.41)

2. Secondary Outcome: Buccolingual Change in Width of Keratinized Soft Tissue
Description: Difference in post operative measurement analysis of keratinized gingiva changes following extraction and alveolar ridge preservation
Time Frame: Soft tissue measurement at time of extraction and grafting and 12 weeks after extraction and grafting
Population: Only nine patients had implants placed within the exact specified 12 week timeframe from the date of extraction, therefore data collection and analysis were only performed on these participants.
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot
Number analyzed (Participants) | 4 | 5
Millimeters | -1 (3.03) | -4 (2.7)

3. Secondary Outcome: Post-operative Pain and Swelling
Description: Post-operative pain and complications measured by VAS-questionnaire obtained following extraction and grafting. The VAS-questionnaire contained the following categories to be answered 7days post-operatively: Pain, Swelling. A visual line scale of 100mm in length was provided with no pain/swelling on the one end and severe pain/swelling on the opposite end. Participants were instructed to rate their pain and swelling by marking a single line on the scale indicating the degree of pain/swelling they experienced. Markings were physically measured on the scale and converted into a score with 0 representing no pain/swelling and 1 representing severe pain/swelling.
Time Frame: Measured at 7 days following extraction and grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot
Number analyzed (Participants) | 14 | 12
score on a scale | 0.22 (0.29) | 0.23 (0.30)

ADVERSE EVENTS:
Time Frame: 12weeks
Description: Patients were monitored 1-2weekly during the 12week healing period and any adverse events recorded by the treating clinician.
Arm/Group | Freeze Dried Bone Allograft | L-PRF Clot
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 7/14 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Freeze Dried Bone Allograft (N=14) | L-PRF Clot (N=12)
Membrane loss earlier than 4weeks (Surgical and medical procedures) | 7 | 3 — Non-resorbable membrane covering the graft material was monitored during healing. Membrane dehiscence or mobility recorded earlier than 4weeks were recorded. Membrane loss did not affect healing or cause infection or loss of the graft.

LIMITATIONS AND CAVEATS:
Initial sample size calculation was 42, due to limited recruitment timeframe and period of study, a limited sample size was obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03331185/Prot_SAP_000.pdf